CLINICAL TRIAL: NCT04902066
Title: Face Your Fears: an Assessor-blinded, RCT Evaluating the Effectiveness of Cognitive Behavioural Virtual Reality Therapy Versus Cognitive Behavioural Therapy in Patients with Schizophrenia Spectrum Disorders.
Brief Title: Face Your Fears: Cognitive Behavioural Virtual Reality Therapy for "Paranoia".
Acronym: FYF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Central Denmark Region (Other); Mental Health Services in the North Denmark Region (Unknown)
Responsible Party: Principal Investigator, Merete Nordentoft, Professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0134-00066B and ID 148727
Record Dates: First submitted 2021-04-19; First posted 2021-05-26 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Paranoid Schizophrenia; Schizophrenia and Related Disorders; Schizophrenia Prodromal; Schizotypal Disorder; Paranoid Ideation; Paranoid Delusion; Ideas of Reference; Psychosis Paranoid; Psychotic Disorders; Psychotic Paranoia; Psychotic; Disorder, Delusional
MeSH Terms: conditions — Schizophrenia, Paranoid; Schizophrenia; Schizotypal Personality Disorder; Paranoid Disorders; Psychotic Disorders; Mental Disorders; Delusions

STUDY DESIGN:
Intervention Model Description: A randomised, assessor-blinded parallel-groups superiority clinical trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Independent assessors blinded to the treatment will evaluate outcome. Investigator's conduct assessment and/or supervise assessments and are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Behavioural Virtual Reality Therapy (CBT-VR) (Experimental): The CBT-VR consists of traditional CBT with the augmentation of virtual reality exposure. The virtual reality exposure comprises four virtual social environments (a bus, café, street, and supermarket). These are daily social situations that generally elicit paranoid thinking in patients with a schizophrenia spectrum disorder. While virtually engaging in these distressing situations, the therapist will facilitate a CBT dialogue aimed at generating alternative (i.e. non-threatening) thinking, diminishing safety behaviours (e.g. social isolation), and building up new coping strategies. This is expected to alleviate distress, anxiety, and improve daily social functioning. Preliminary findings reveal this virtual reality program to be well-tolerated and highly effective in reducing paranoia and anxiety in psychosis. Patients will be offered 10 individual sessions.
  Interventions: Other: Cognitive Behavioural Virtual Reality Therapy.
- Traditional Cognitive Behavioural Therapy (Active Comparator): The treatment in the CBT group will follow the core principles of CBT used for psychotic disorders. The CBT treatment facilitates an individualised, problem-oriented approach, and uses key CBT techniques such as developing a problem and goal list, normalising psychotic-like experiences, evaluation of appraisals, and removing or diminishing safety behaviour. Patients will be offered 10 individual sessions.
  Interventions: Other: Traditional Cognitive Behavioural Therapy

INTERVENTIONS:
Other: Cognitive Behavioural Virtual Reality Therapy. — Cognitive Behavioural Therapy augmented with Virtual Reality.
  Arms: Cognitive Behavioural Virtual Reality Therapy (CBT-VR)
Other: Traditional Cognitive Behavioural Therapy — Traditional Cognitive Behavioural Therapy for psychosis.
  Arms: Traditional Cognitive Behavioural Therapy

SUMMARY:
The study is a randomised, assessor-blinded parallel-groups superiority clinical trial fulfilling the CONSORT criteria for non-pharmacological treatment. A total of 256 patients will be allocated to either Cognitive Behavioural Virtual Reality Therapy plus treatment as usual, versus traditional CBT for psychosis plus treatment as usual. All participants will be assessed at baseline and 3- and 9 months post baseline. A stratified block-randomisation with concealed randomisation sequence will be conducted. Independent assessors blinded to the treatment will evaluate outcome. Analysis of outcome will be carried out with the intention to treat principles.

DETAILED DESCRIPTION:
Ideas of reference and ideas of persecution are among the most frequent symptoms in psychotic disorders, and they hinder patients in conducting daily activities such as leaving the home or using public transportation - as well as inflicting immensely on their quality of life. The social avoidance caused by these symptoms does not improve with antipsychotic mediation. Cognitive behavioural therapy (CBT) for psychosis has demonstrated beneficial effect on psychotic symptoms, but the average effect sizes are in the small to moderate range, and training and resource requirements mean that, in practice, therapy is not delivered to all those who might benefit. Hence, there is considerable interest in the development of novel therapies that draw on the principles of cognitive behavioural therapy for psychosis, but which are shorter, more effective, and are capable of being delivered by a wider workforce. Augmenting CBT with virtual reality exposure has the possibility of creating artificial experiences in real time, that make the user feel immersed and able to interact as if it was the real world. Additionally, virtual reality therapy allows for personalization of the therapy to match the specific social challenges of each patient. Preliminary findings suggest virtual reality exposure to lead to faster symptom reduction than traditional therapy. While the potential beneficial effects of virtual reality exposure to psychotic, and sub-threshold psychotic symptoms, such as ideas of reference and ideas of persecution, are evident and virtual reality therapies are promising in general, the research field is in an urgent need of evidence on the effectiveness of virtual reality therapy in patients with schizophrenia spectrum disorders. The proposed trial is hitherto the largest trial in the world to evaluate the effectiveness of cognitive behavioural virtual reality therapy (CBT-VR) compared to traditional CBT. The investigators expect to find CBT-VR to be more beneficial in reducing ideas of reference and ideas of persecution in patients with schizophrenia spectrum disorders. Additionally, the investigators expect it to result in improved depressive, anxiety-, and negative symptoms, as well as improved social cognition and psychosocial functioning and quality of life in patients with schizophrenia spectrum disorders. The target group in the trial also encompass patients with schizotypal disorder (often young adults), showing subthreshold psychotic symptoms (e.g. ideas of reference), that are at increased risk of developing manifest psychosis. The CBT-VR may show efficacy in preventing progression to an overt psychotic state in these patients. Hence, there is a great potential for CBT-VR in the treatment of patients with psychosis and sub-threshold psychosis, but studies are needed to establish evidence for the treatment. If the results of the current trial are positive, the manualised treatment can easily be implemented in clinical practise.

Note:

When the trial was initiated, the original primary outcome was ideas of persecution, measured with part B in Green Paranoid Thought Scale (GPTS) while ideas of social reference, measured with part A in Green Paranoid Thought Scale, was listed as a secondary outcome in the trial protocol, here on Clinicaltrials.gov and in the approval from the Committee on Health Research Ethics of the Capital Region Denmark.

During our trial, our impressions in the clinical assessments were, that ideas of social reference seem to be a more appropriate primary outcome due to our population including people diagnosed with schizotypal disorders along with participants with manifest psychotic disorders.

We observed that participants with schizotypal disorders experiencing ideas of social reference, that are more attenuated paranoid ideations, would often receive a low score on the GPTS part B. Therefore, listing GPTS part B as primary outcome would hypothetically only reflect the symptom level of part of the study population (patients with manifest psychosis), while not fully comprising the symptom level, and potential for change, found in the population of patients with schizotypal disorder. ''

As of February, 23 2022, 10 months into the trial, where 79 participants out of 256 were included and had participated in baseline assessments, we decided after thorough consideration to exchange our primary outcome, GPTS part B, ideas of persecution, with our secondary outcome, GPTS part A, ideas of social reference, as this was intended to capture the symptom level in the total study population.

The exchange did not affect participation in our trial or the informed consent. Intervention in both groups and measurements were unchanged. The two outcomes constitute together GPTS and the unifying concept we attempt to treat, namely paranoid ideations. As this is a blinded, methodologically sound trial, we had not (and still have not throughout the study period) access to preliminary data and therefore no knowledge of the distribution of our two intervention groups nor the potential effect of the intervention.

The power calculation remains unchanged irrespective of the selection of primary outcome. (Ideas of persecution: relevant difference 6.0, SD 17.9, N=128*2, power= 80%). Due to the notions mentioned above, we did not find any reasons for ethical implications of the change of primary outcome - as we also were fully transparent with this change of outcome here on Clinicaltrials.gov.

We therefore assumed that our ethical committee would approve of this change. However, on September 3 2022 we received a rejection from the Committee on Health Research Ethics of the Capital Region Denmark on changing outcomes, on the invariable grounds that the trial is commenced. This means that it is necessary to keep ideas of persecution, part B in Green Paranoid Thought Scale, as our primary outcome and keep ideas of social reference, part A in Green Paranoid Thought Scale as a secondary outcome.

A design paper was published while we had ideas of social reference, part A in Green Paranoid Thought Scale, as a primary outcome. An Update, informing about this significant change in the form of changing back to the originally, approved, primary outcome, has been published.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - years
2. Ability to give informed consent
3. A schizophrenia spectrum disorder (ICD-10 code: F20 -F29)
4. Green Paranoid Thought Scale total score ≥ 40

Exclusion Criteria:

1. Rejecting informed consent
2. A diagnosis of organic brain disease
3. IQ of 70 or lower (known mental retardation as assessed by medical record)
4. A command of spoken Danish or English inadequate for engaging in therapy
5. Inability to tolerate the assessment process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 254 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
(GPTS) Green Paranoid Thought Scale Part B: Ideas of persecution. | 3 months from inclusion
  The primary outcome is level of ideas of persecution measured with Green Paranoid Thought Scale at cessation of treatment at 3-months. The Green Paranoid Thought Scale has displayed good reliability and validity in patients with psychosis, displaying paranoid, persecutory delusions, and has also been used in patients at-risk for psychosis showing subthreshold psychotic symptoms.
  Minimum total score: 32. Maximum total score: 160. Part A (Ideas of social reference) minimum score: 16 and maximum score: 80. Part B (ideas of persecution) minimum score 16 and maximum score: 80. Part B score = or > 45 are assumed to be threshold for development of persecutory delusion.
  Higher score means worse outcome.

SECONDARY OUTCOMES:
SIAS (Social Interaction Anxiety Scale) | 3 and 9 months from inclusion
  Minimum score: 0 Maximum score: 20*4=80. Item 5,9 and 11 have reverse score. Higher score means worse outcome.
SBQ (Safety Behaviour Questionnaire) | 3 and 9 months from inclusion
  Minimum score: 0. Maximum score is in theory unlimited depending on the number of identified, specific safety behaviours.
PSP (Personal and Social Performance Scale) | 3 and 9 months from inclusion
  Minimum score: 1 Maximum score: 100. Higher score means better outcome.
CANTAB ERT (Emotion Recognition Task) | 3 and 9 months from inclusion
(GPTS) Green Paranoid Thought Scale Part A: Ideas of social reference | 3 and 9 months from inclusion
  Minimum total score: 32. Maximum total score: 160. Part A (Ideas of social reference) minimum score: 16 and maximum score: 80. Part B (Ideas of persecution) minimum score 16 and maximum score: 80. Part B score = or > 45 are assumed to be threshold for development of delusion. Higher score means worse outcome.
(GPTS) Green Paranoid Thought Scale Part B: Ideas of persecution | 9 months from inclusion
  Minimum total score: 32. Maximum total score: 160. Part A (Ideas of social reference) minimum score: 16 and maximum score: 80. Part B (Ideas of persecution) minimum score 16 and maximum score: 80. Part B score = or > 45 are assumed to be threshold for development of delusion. Higher score means worse outcome.

OTHER OUTCOMES:
CDSS (Calgary Depression Scale for Schizophrenia) | 3 and 9 months from inclusion
  Minimum score: 0 Maximum score: 9*3 = 27. Higher score means worse outcome.
BNSS (Brief Negative Symptom Scale) | 3 and 9 months from inclusion
  13 items with a score from minimum 0 to maximum 6 for each item. Higher score means worse outcome.
COGDIS (Cognitive disturbances scale) | 3 and 9 months from inclusion
  Score of 0-6 indicate a range. Minimum score: 0 Maximum score: 9*6 = 54. Higher score means worse outcome. Trait phenomenons are coded with a "7", unknown degree of severly is coded with a "8" and uncertainty whether the symptom is present is coded with a "9".
SAPS (Scale for the Assesment of Positive symptoms) | 3 and 9 months from inclusion
  Composite total score: Minimum score: 0 Maximum score: 30*5 = 150. Higher score means worse outcome.
  Global score: Minimum score: 0 Maximum score: 4*5 = 20. Higher score means worse outcome.
Trustworthiness Scale | 3 and 9 months from inclusion
  Minimum score: -3*42=-126 Maximun score: +3*42=126. Higher positive score means better outcome. Higher negative score means worse outcome.
DACOBS (Davos Assessment of the Cognitive Biases Scale) | 3 and 9 months from inclusion
  Total score: Minimum score: 1*42=42. Maximum score:7*42=294. Higher score means worse outcome.
  Subscales of:
  Jumping to conclusions bias: Item 3+8+16+18+25+30 Belief Inflexibility bias: Item 13+15+26+34+38+41 Attention for Threat bias: Item 1+2+6+10+20+37 External Attribution bias: Item 7+12+17+22+24+29
  Social Cognition problems: Item 4+9+11+14+19+39 Subjective Cognitive problems: Item 5+21+28+32+36+40
  Safety behaviors: Item 23+27+31+33+35+42
SIDAS (Suicidal Ideation Attributes Scale) | 3 and 9 months from inclusion
  Minimum score: 0. Maximum score: 50. Item 2 has a reverse score. Higher score means worse outcome.
BCSS (The Brief Core Schema Scales: Beliefs about self and others) | 3 and 9 months from inclusion
  Items with negative belief of self and others: Minimum score: 0. Maximum score: 2*6*4= 48. Higher score means worse outcome.
  Items with Positive belief of self and others: Minimum score: 0. Maximum score: 2*6*4= 48. Higher score means better outcome.
SSPA (Social Skills Performance Assessment) | 3 and 9 months from inclusion
  Scene I: Minimum score: 1*8=8. Maximum score: 5*8:40. Higher score means better outcome.
  Scene II: Minimum score: 1*9=9. Maximum score: 5*9:45. Higher score means better outcome.
TALE (Trauma And Life Events checklist) | Baseline measure
IBT (Intentionality Bias Task) | 3 and 9 months from inclusion
(R-GPTS) Revised Green Paranoid Thought Scale | 3 and 9 months from inclusion
  Minimum total score: 0. Maximum total score: 4*18=72. Part A (Ideas of social reference) minimum score: 0 and maximum score: 4*8=32. Part B (Ideas of persecution) minimum score 0 and maximum score: 4*10=40. Part B score = or > 18 are assumed to be threshold for development of delusion. Higher score means worse outcome.
GSE (General Self Efficacy Scale) | 3 and 9 months from inclusion
  Minimum score: 1*10=10. Maximum score: 4*10=40. Higher score means better outcome.
Big-5 (personality traits) | 3 and 9 months from inclusion
  5 spectrums of personality traits assessed with 5 items each.
  Minimum score for each personality trait: Minimum score: 1*5=5. Maximum score: 5*5=25
  Certain items have reverse scores.
EQ-5D-5L (EuroQOL five dimensions questionnaire) | 3 and 9 months from inclusion
  Scoring the descriptive system:
  Minimum score: 1-1-1-1-1. Maximum score: 5-5-5-5-5. Higher score means worse outcome.
  Scoring the VAS:
  Minimum score: 0. Maximum score: 100. Higher score means better outcome.
WHO (World Health Organization 5) | 3 and 9 months from inclusion
  Minimum score: 0. Maximum score: 5*5*4=100. Higher score means better outcome.
CSQ (Client Satisfaction Questionnaire) | 3 months follow-up
SFS (The Social Functioning Scale) | 3 and 9 months from inclusion
  Minimum raw score: 0. Maximum raw score: 15+9+39+45+66+39+19=223. Higher score means better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Research Center for Mental Health - CORE, Copenhagen, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeppesen UN, Vernal DL, Due AS, Mariegaard LS, Pinkham AE, Austin SF, Vos M, Christensen MJ, Hansen NK, Smith LC, Hjorthoj C, Veling W, Nordentoft M, Glenthoj LB. Virtual reality-based versus standard cognitive behavioral therapy for paranoia in schizophrenia spectrum disorders: a randomized controlled trial. Nat Med. 2025 Oct;31(10):3425-3439. doi: 10.1038/s41591-025-03880-8. Epub 2025 Aug 13. PMID 40804323
- [Derived] Jeppesen UN, Due AS, Mariegaard L, Pinkham A, Vos M, Veling W, Nordentoft M, Glenthoj LB. Update to the study protocol Face Your Fears: Virtual reality-based cognitive behavioral therapy (VR-CBT) versus standard CBT for paranoid ideations in patients with schizophrenia spectrum disorders: a randomized clinical trial. Trials. 2023 Jan 23;24(1):52. doi: 10.1186/s13063-023-07069-7. PMID 36691039
- [Derived] Jeppesen UN, Due AS, Mariegaard L, Pinkham A, Vos M, Veling W, Nordentoft M, Glenthoj LB. Face Your Fears: Virtual reality-based cognitive behavioral therapy (VR-CBT) versus standard CBT for paranoid ideations in patients with schizophrenia spectrum disorders: a randomized clinical trial. Trials. 2022 Aug 15;23(1):658. doi: 10.1186/s13063-022-06614-0. PMID 35971137